CLINICAL TRIAL: NCT00268489
Title: A Phase II Study of Pemetrexed Disodium (ALIMTA®) Plus Bevacizumab in Patients With Stage IIIB Pleural Effusion or Stage IV Non-Small Cell Lung Cancer (Second-Line Treatment)
Brief Title: Pemetrexed Disodium and Bevacizumab in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0426; NCI-2012-02681 (Registry Identifier: CTRP (Clinical Trials Reporting System)); SWOG-N0426; CDR0000456427 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Bevacizumab; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pemetrexed + bevacizumab (Experimental): Patients receive pemetrexed disodium IV over 10 minutes and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  After completion of study treatment, patients are followed periodically for 5 years.
  Interventions: Biological: bevacizumab; Drug: pemetrexed disodium

INTERVENTIONS:
Biological: bevacizumab
Drug: pemetrexed disodium

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as pemetrexed disodium, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving pemetrexed disodium together with bevacizumab may be an effective treatment for non-small cell lung cancer.

PURPOSE: This phase II trial is studying how well giving pemetrexed disodium together with bevacizumab works in treating patients with stage III or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the 3 month progression-free survival rate of the combination of pemetrexed disodium with bevacizumab in a patient population with stage IIIB (due to pleural effusion) or IV non-small cell lung cancer.

Secondary

* Determine the tumor response rate in these patients.
* Determine the effect of pemetrexed disodium in combination with bevacizumab on overall survival and duration of response in these patients.
* Determine the toxicity profile of this drug regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive pemetrexed disodium IV over 10 minutes and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically diagnosed stage IIIB or IV non-small cell lung cancer

  * Stage IIIB patients must have pleural effusion

    * No symptomatic serosal effusion (grade 2 dyspnea) that is not amenable to drainage
  * Mixed histology allowed if all components consistent with non-small cell lung cancer
  * Tumors with squamous cell histology feature are allowed
* Must have measurable disease with at least one lesion with a longest diameter accurately measured as ≥ 2.0 cm with conventional techniques or as ≥ 1.0 cm with spiral CT

  * Large ( > 4 cm) centrally located lesions or large lesions in close proximity to major blood vessels should receive palliative radiation

    * The irradiated lesion should not be a target lesion
* Previously treated with one chemotherapy regimen in the neoadjuvant, adjuvant, or advanced disease setting
* No symptomatic, untreated, or uncontrolled CNS metastases

  * CNS metastases treated with prior whole brain radiotherapy allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/ mm^3
* Hemoglobin ≥ 9 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN) or direct bilirubin normal
* AST and ALT ≤ 3 times ULN (5 times ULN if liver has tumor involvement)
* Creatinine clearance ≥ 45 mL/min
* Urine protein:creatinine ratio < 1.0
* Pregnant or nursing women are ineligible
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No seizure disorder
* No clinically significant infection
* No other second primary malignancy within the past 5 years except carcinoma in situ of the cervix, non-melanomatous skin cancer, or low-grade (Gleason score ≤ 6) localized prostate cancer
* No hypertension or labile hypertension
* No history of poor compliance with antihypertensive medications
* No angina pectoris
* No congestive heart failure within the past 3 months unless ejection fraction > 40%
* No myocardial infarction within the past 6 months
* No cardiac arrhythmia
* No interstitial pneumonia or extensive and symptomatic interstitial fibrosis of the lung
* No active or recent history of hemoptysis

  * Hemoptysis resolved > 2 weeks ago with measures such as palliative radiation therapy (i.e., 3,000 cGy over 10 fractions), arteriographic embolization, or endobronchial interventions (e.g., photodynamic therapy or brachytherapy) is acceptable
* No diabetes
* No prior serious, non-healing wounds, ulcers, or bone fractures
* No history of stroke within the past 6 months
* No history of abdominal fistula or gastrointestinal perforation
* No intra-abdominal abscess within the past 6 months
* Not at greater than average risk of bleeding
* No significant traumatic injury within the past 4 weeks

PRIOR CONCURRENT THERAPY:

* No aspirin at doses ≥ 1.3 grams per day within 10 days prior to or 10 days after pemetrexed disodium treatment
* No chemotherapy within the past 3 weeks (6 weeks for mitomycin C or nitrosoureas)
* No immunotherapy or biologic therapy within the past 2 weeks
* No full field radiation therapy within the past 4 weeks or limited field radiation therapy within the past 2 weeks

  * The site of previous radiotherapy should have evidence of progressive disease if it is the only site of disease
* No prior post pelvic radiation
* No prior use of pemetrexed disodium
* No prior radiation to > 25% of the marrow cavity
* No major surgery (i.e., laparotomy) or open biopsy within the past 4 weeks
* No minor surgery within the past 2 weeks except insertion of a vascular access device
* No concurrent major surgery
* No other chemotherapy, immunotherapy, hormonal therapy, radiotherapy, or any ancillary therapy considered investigational within the past 4 weeks
* No concurrent use of Hypericum perforatum (St. John's wort)
* No concurrent anticoagulant use

  * Low-dose warfarin or heparin for deep venous thrombosis prophylaxis allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-05; Primary Completion 2007-05 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Proportion of progression-free patients at 3 months | at 3 months

SECONDARY OUTCOMES:
Response (complete and partial) as assessed by RECIST criteria | Up to 5 years
Overall survival | Up to 5 years
Progression-free survival | Up to 5 years
Duration of response | Up to 5 years
Time to treatment failure | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alex A. Adjei, MD, PhD, Study Chair — Roswell Park Cancer Institute
Locations (248):
- United States (248):
  - Providence Cancer Center, Anchorage, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Eden Medical Center, Castro Valley, California
  - Saint Rose Hospital, Hayward, California
  - Highland General Hospital at St. George's University School of Medicine, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Ted B. Wahby Cancer Center at Mount Clemens General Hospital, Mount Clemens, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA at Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Adjei AA, Mandrekar SJ, Dy GK, Molina JR, Adjei AA, Gandara DR, Ziegler KL, Stella PJ, Rowland KM Jr, Schild SE, Zinner RG. Phase II trial of pemetrexed plus bevacizumab for second-line therapy of patients with advanced non-small-cell lung cancer: NCCTG and SWOG study N0426. J Clin Oncol. 2010 Feb 1;28(4):614-9. doi: 10.1200/JCO.2009.23.6406. Epub 2009 Oct 19. PMID 19841321
- [Result] Adjei AA, Mandrekar SJ, Dy GK, et al.: A phase II second-line study of pemetrexed (pem) in combination with bevacizumab (bev) in patients with advanced non-small cell lung cancer (NSCLC): An NCCTG and SWOG study. [Abstract] J Clin Oncol 26 (Suppl 15): A-8080, 2008.